CLINICAL TRIAL: NCT01380392
Title: The Illness of Uncertainty, Personality and Coping Strategies in Patients With Hepatocellular Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Shiow-Ching Shun, Department of Nursing,NTU
Other Study IDs: 201101063RC
Record Dates: First submitted 2011-06-22; First posted 2011-06-27 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Liver Carcinoma
Keywords: Liver cancer; Uncertainty; Personality; coping strategies
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The aims of this study are to (1) understand the uncertainty , personality and coping strategies in patients with HCC, and identify the significant factors for coping.

DETAILED DESCRIPTION:
A cross-sectional correlated design will be used and (2) patients will be recruited by purposive sampling from wards and outpatient departments at a medical center in Taipei.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Has HCC and knows condition
* Con's clear
* Agree join the study

Exclusion Criteria:e

* BCLC stage C or D
* Accepted C/T, R/T,target therapy or supportive care
* Patient who receive liver transplantation

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HCC patients who accept surgical or medical treatment.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-02; Primary Completion 2012-02 (Estimated); Study Completion 2012-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Shiow-Ching Shun, Doctor, Study Chair — National Taiwan University
Locations (1):
- Research Nurse, Taipei, Taiwan